CLINICAL TRIAL: NCT06065553
Title: Study on the Prevalence of Psychiatric and Substance Abuse Disorders Among People in Precarious Situations, Extreme Exclusion and/or Wandering on Cayenne and Its Surroundings.
Brief Title: Prevalence of Psychiatric and Substance Abuse Disorders Among People in Precarious Situations in Cayenne
Acronym: EPICEA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: EPICEA
Record Dates: First submitted 2023-06-07; First posted 2023-10-04 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Psychiatric Disorder; Substance Use Disorders
Keywords: Psychiatric disorders; Substance abuse; Precarity; French Guiana
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, descriptive, cross-sectional, single-center study. The main objective of the study is to estimate the prevalence of the main psychiatric disorders and substance abuse disorders among people living in precarious, excluded and/or wandering on Cayenne and its surroundings

DETAILED DESCRIPTION:
In French Guiana, the mental health care and support system (health, medical-social, social, associative and institutional structures) is structurally lagging behind.

The density of specialist professionals is low; the psychiatric private sector is absent.

In order to adapt care provision, it is necessary to gain a better understanding of certain target populations, in particular those with multiple vulnerabilities, who have specific needs and expectations.

As highlighted by the results of a number of studies already carried out in France and elsewhere in the world, psychaitric disorders and substance-related addictive disorders have a greater impact on people living in situations of extreme exclusion, precariousness and homelessness.

In 2017, in French Guiana, one person out of two lives below the poverty line, compared to 14.9% in France.

A recent study estimated the prevalence rate of psychiatric disorders in the general population of the CACL (Communauté d'Agglomération du Centre Littoral) in French Guiana (SMPG - Santé Mentale en Population générale - study in 2021). Nowadays, there is no recent study measuring the prevalence of psychiatric disorders specifically among populations in precarious situations, wandering and/or extreme exclusion on Cayenne Island.

The main hypothesis of the research would therefore be to observe a prevalence of psychiatric disorders and addictive disorders in the precarious population that is at least as high, if not higher, than in the general population of the CACL.

Another hypothesis of the research would be to find that the distribution of the prevalence of each psychiatric disorder is not identical to that found in the general population of the CACL (more addictive disorders and more psychotic disorders in the precarious population, more disorders linked to post-traumatic stress disorder in migrant populations).

Another research hypothesis would be to observe that the use of healthcare and the perception of health are different from those of the general population of the CACL, and that it is therefore necessary to develop appropriate human and structural resources.

However, it seems essential to know this prevalence in order to adjust the offer of care and adapt it as much as possible to the specific needs of this population.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* person who uses support services intended for people in situations of precariousness, extreme exclusion and/or wandering on Cayenne and its surroundings - person agreeing to participate in the study.

Exclusion Criteria:

* Person refusing to participate in the study
* Person presenting an acute state of decompensation of a psychiatric pathology and/or a state of crisis (agitation crisis, suicidal crisis) and/or confusion or presenting an acute intoxication to a substance preventing him/her from understanding and answering questions.
* Impossibility of having an interpreter for a person with no (or little) French

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in precarious situations, extreme exclusion and/or wandering on Cayenne and its surroundings
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychiatric disorders and substance abuse disorders | Baseline
  To estimate the prevalence of the main psychiatric disorders, as well as the prevalence of addictive disorders to psychoactive substances among people in a precarious situation, excluded and/or wandering on Cayenne Island and who use primary care services

SECONDARY OUTCOMES:
Description of socio-demographic profiles | Baseline
  Describe the different socio-demographic profiles of people in a precarious situation, excluded and/or wandering on Cayenne Island and who use primary care services.
Description of perceived health status | Baseline
  To describe the perceived health status of people in a precarious situation, excluded and/or wandering on Cayenne Island and who use primary care services
Description of use and access to health care | Baseline
  To describe the use of and access to care for people in a precarious situation, excluded and/or wandering on Cayenne Island and who use primary care services

CONTACTS AND LOCATIONS:
Overall Officials: Caroline JANVIER, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hossain MM, Sultana A, Tasnim S, Fan Q, Ma P, McKyer ELJ, Purohit N. Prevalence of mental disorders among people who are homeless: An umbrella review. Int J Soc Psychiatry. 2020 Sep;66(6):528-541. doi: 10.1177/0020764020924689. Epub 2020 May 28. PMID 32460590
- [Background] Ayano G, Shumet S, Tesfaw G, Tsegay L. A systematic review and meta-analysis of the prevalence of bipolar disorder among homeless people. BMC Public Health. 2020 Jun 9;20(1):731. doi: 10.1186/s12889-020-08819-x. PMID 32513264
- [Background] Ayano G, Solomon M, Tsegay L, Yohannes K, Abraha M. A Systematic Review and Meta-Analysis of the Prevalence of Post-Traumatic Stress Disorder among Homeless People. Psychiatr Q. 2020 Dec;91(4):949-963. doi: 10.1007/s11126-020-09746-1. PMID 32415465
- [Background] Ayano G, Tesfaw G, Shumet S. The prevalence of schizophrenia and other psychotic disorders among homeless people: a systematic review and meta-analysis. BMC Psychiatry. 2019 Nov 27;19(1):370. doi: 10.1186/s12888-019-2361-7. PMID 31775786
- [Background] Fazel S, Geddes JR, Kushel M. The health of homeless people in high-income countries: descriptive epidemiology, health consequences, and clinical and policy recommendations. Lancet. 2014 Oct 25;384(9953):1529-40. doi: 10.1016/S0140-6736(14)61132-6. PMID 25390578
- See also: Mental health status of homeless people in Paris, 1997 — https://bdoc.ofdt.fr/index.php?lvl=notice_display&id=59199
- See also: Mental health status and abuse disorders of homeless people in Paris region, 2010 — https://www.inserm.fr/wp-content/uploads/2017-11/inserm-rapportthematique-sementa-2010.pdf
- See also: When homelessness puts at risk children mental health — https://www.samusocial.paris/sites/default/files/2022-11/HD_WEB_Synthese_SAMU_pageapage.pdf
- See also: Public Health Aspects of Mental Health Among Migrants and Refugees: A Review of the Evidence on Mental Health Care for Refugees, Asylum Seekers and Irregular Migrants in the WHO European Region — https://www.ncbi.nlm.nih.gov/books/NBK391045/
- See also: Health survey in French Overseas department — https://www.santepubliquefrance.fr/etudes-et-enquetes/barometres-de-sante-publique-france/barometre-sante-dom-2014
- See also: MINI questionnaire — https://www.researchgate.net/publication/280880465_Mini_International_Neuropsychiatric_Interview_French_current_DSM-IV
- See also: PTSD screen for DSM-5 — https://www.ptsd.va.gov/professional/assessment/screens/pc-ptsd.asp